CLINICAL TRIAL: NCT04994691
Title: Effect of Varied Outreach Methods on Appointment Scheduling and Appointment Completion Using MyChart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020-0769-2
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — NMT1 protein, S pombe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No message (Placebo Comparator): No message sent
  Interventions: Other: No Message
- Standard message (Active Comparator): 2 MyChart reminders that child is overdue for well child check visit
  Interventions: Other: Standard message
- Tailored message (Active Comparator): 2 MyChart reminders that child is overdue for well child check visit with date of last WCC and age
  Interventions: Other: Tailored message

INTERVENTIONS:
Other: No Message — No messages are sent
  Arms: No message
Other: Standard message — 2 MyChart reminders that child is overdue for well child check visit
  Arms: Standard message
Other: Tailored message — 2 MyChart reminders that child is overdue for well child check visit with date of last WCC and age
  Arms: Tailored message

SUMMARY:
Our objective is to determine the effectiveness of varied outreach methods (e.g. standard versus tailored MyChart messaging) to children age 6-17 years old who are due for a WCC visit and don't have one scheduled in the next 45 days on the outcomes of appointment scheduling and appointment completion.

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years
* has not had a well child check in past 365 days
* no future well child check visit scheduled
* parent preferred language = English or Spanish

Exclusion Criteria:

* no active MyChart account

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 945 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berset AE, Burkhardt MC, Xu Y, Mescher A, Brinkman WB. Effect of Electronic Outreach Using Patient Portal Messages on Well Child Care Visit Completion: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242853. doi: 10.1001/jamanetworkopen.2022.42853. PMID 36399342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Message | Standard Message | Tailored Message
Started | 315 | 315 | 315
Completed | 315 | 315 | 315
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Message | Standard Message | Tailored Message | Total
Number analyzed (Participants) | 315 | 315 | 315 | 945
Age, Customized [Count of Participants; unit: Participants]
  6-8y | 137 | 133 | 134 | 404
  9-11y | 96 | 98 | 98 | 292
  12-14y | 33 | 40 | 38 | 111
  15-17y | 49 | 44 | 45 | 138
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 152 | 167 | 493
  Male | 141 | 163 | 148 | 452
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American Non-Hispanic | 211 | 184 | 195 | 590
  White Non-Hispanic | 71 | 82 | 73 | 226
  Multiracial Non-Hispanic | 15 | 21 | 15 | 51
  Missing Data Hispanic | 5 | 6 | 11 | 22
  Asian Non-Hispanic | 5 | 10 | 4 | 19
  White Hispanic | 3 | 5 | 10 | 18
  Missing Data Non-Hispanic | 1 | 3 | 3 | 7
  Black or African American Hispanic | 2 | 3 | 1 | 6
  Multiracial Hispanic | 1 | 1 | 1 | 3
  American Indian and Alaska Native Non-Hispanic | 0 | 0 | 1 | 1
  Middle Eastern Non-Hispanic | 0 | 0 | 1 | 1
  Native Hawaiian and Other Pacific Islander Hispanic | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Well Child Check Visit
Description: Participants completed well child check visit as determined by presence of a well visit billing code documentation in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 315 | 315 | 315
Participants | 40 | 76 | 61
Statistical Analysis 1: Comparison: No Message vs Standard Message; Test type: Superiority; p = 0.000, Regression, Logistic; Risk Ratio (RR) = 1.92, 95% CI 2-sided [1.38 to 2.60] — Standard Message vs. No Message
Statistical Analysis 2: Comparison: No Message vs Tailored Message; Test type: Superiority; p = 0.023, Regression, Logistic; Risk Ratio (RR) = 1.52, 95% CI 2-sided [1.06 to 2.13] — Tailored Message vs. No Message
Statistical Analysis 3: Comparison: Standard Message vs Tailored Message; Test type: Superiority; p = 0.124, Regression, Logistic; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.94 to 1.66] — Standard Message vs. Tailored Message

2. Secondary Outcome: Number of Participants Who Scheduled an Appointment for a Well Child Check Visit.
Description: Participant scheduled a well child check visit as determined by electronic health record documentation.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 315 | 315 | 315
Participants | 30 | 58 | 47
Statistical Analysis 1: Comparison: No Message vs Standard Message; Test type: Superiority; p = 0.001, Regression, Logistic; Risk Ratio (RR) = 1.97, 95% CI 2-sided [1.32 to 2.84] — Standard Message vs. No Message
Statistical Analysis 2: Comparison: No Message vs Tailored Message; Test type: Superiority; p = 0.040, Regression, Logistic; Risk Ratio (RR) = 1.57, 95% CI 2-sided [1.02 to 2.34] — Tailored Message vs. No Message
Statistical Analysis 3: Comparison: Standard Message vs Tailored Message; Test type: Superiority; p = 0.202, Regression, Logistic; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.88 to 1.74] — Standard Message vs. Tailored Message

3. Secondary Outcome: Number of Participants Who Received Their First COVID-19 Vaccination
Description: Participant receipt of their first COVID-19 vaccination as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of the intervention or the date of randomization for the control group
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 82 | 84 | 83
Participants | 3 | 14 | 4

4. Post Hoc Outcome: Number of Participants Who Received DTaP Vaccination
Description: Participant receipt of DTaP vaccination as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Population: Analysis includes all patients eligible to receive this vaccine during the 8-week study period
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 32 | 32 | 34
Participants | 8 | 6 | 6

5. Post Hoc Outcome: Number of Participants Who Received HPV Vaccination
Description: Participant receipt of HPV vaccination as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Population: Analysis includes all patients eligible to receive this vaccine during the 8-week study period
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 50 | 49 | 52
Participants | 7 | 13 | 9

6. Post Hoc Outcome: Number of Participants Who Received MCV4 Vaccination
Description: Participant receipt of MCV4 vaccination as determined by presence of documentation of vaccine administration in the electronic health record.
Time Frame: Within 8 weeks of the date of intervention or the date of randomization for the control group
Population: Analysis includes all patients eligible to receive this vaccine during the 8-week study period
Measure: Count of Participants; unit: Participants
Arm/Group | No Message | Standard Message | Tailored Message
Number analyzed (Participants) | 49 | 54 | 57
Participants | 9 | 10 | 12

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | No Message | Standard Message | Tailored Message
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/315 | 0/315
Serious Adverse Events (participants affected / at risk) | 0/315 | 0/315 | 0/315
Other Adverse Events (participants affected / at risk) | 0/315 | 0/315 | 0/315

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT04994691/Prot_SAP_000.pdf